CLINICAL TRIAL: NCT05034263
Title: Imaging a Cholinergic Biomarker of Cognition in Parkinson's Disease
Status: Terminated | Type: Observational
Why Stopped: Discontinuation of funding.
Sponsor: Stony Brook University (Other)
Collaborators: Parkinson's Foundation (Other)
Responsible Party: Principal Investigator, Chuan Huang, Assistant Professor of Radiology, Stony Brook University
Other Study IDs: 2020-00669
Record Dates: First submitted 2021-08-17; First posted 2021-09-05 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease
Keywords: Acetylcholine; PET; MRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an imaging study designed to illuminate the function of the cholinergic system and its association with cognitive skills in people with Parkinson's disease. The hypothesis of this study is that there will be an association between cholinergic terminal density, sex hormones, and cognitive functioning. Participants will receive a PET and MRI scan along with a battery of neurocognitive tests at baseline and again at 18 months follow-up. Hormone levels will be measured at baseline.

DETAILED DESCRIPTION:
This is an imaging study designed to illuminate the functioning of the cholinergic system in people with Parkinson's disease. Some people with Parkinson's disease develop trouble with certain aspects of thinking such as memory. Studies have shown an association between a decline in thinking skills and dysfunction of the cholinergic system. This study will use the novel PET tracer [18F]VAT to provide more specific information about how the cholinergic system works by enabling direct measurement of cholinergic terminal density and projections. The hypothesis of this study is that there will be an association between cholinergic terminal density, sex hormones, and cognitive functioning. This is a longitudinal observational study that involves a screening visit and four study visits over the course of 18 months. The visits consist of neurocognitive assessments and imaging (MRI and PET scans) administered at baseline and at 18 months follow-up. Hormone levels will also be measured at baseline. This study is open to people with Parkinson's disease who have either normal cognition or mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80
* Diagnosis of Parkinson's disease
* Ability to provide informed consent
* Ability to speak English
* Normal cognition or mild cognitive impairment
* Willingness to go off parkinsonian medication for 12 hours prior to two of the study visits

Exclusion Criteria:

* Contraindication for MRI
* Abnormal clinical brain MRI, specifically with evidence of large-vessel stroke or mass lesion
* History of stereotactic or ablative brain surgery
* Pregnancy
* Recent participation in other research studies involving radiation such that the annual research radiation dose would exceed FDA Limit if participating in this study
* Prior brain injury (eg., TBI)
* Baseline cognitive impairment due to genetic or developmental disorder
* Active illicit drug use or alcohol abuse
* Incapable of staying still for a 2-hour PET or MRI study
* Use of CNS-penetrating medications affecting the cholinergic system, including cholinesterase inhibitors and anticholinergics, up to 60 days prior to study participation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's disease who have normal cognition or mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Cholinergic terminal density at baseline | Baseline
  Measured by PET scan 18F[VAT] distribution volume
Cholinergic terminal density change between baseline and 18-months follow-up | Baseline and 18 months follow-up
  Measured by the difference in PET scan 18F[VAT] distribution volume at baseline and 18-months follow-up
Overall cognitive functioning at baseline | Baseline
  As measured by the Montreal Cognitive Assessment (MoCA). The MoCA measures eight domains commonly affected by mild cognitive impairment. The one-page 30-point test includes assessments of short-term and delayed memory recall, visuospatial abilities, language, orientation to time and space, and executive functions including attention, concentration, and working memory. The MoCA has been shown to be sensitive to change over time. Scores on the MocA range from 0-30 with higher scores indicating better cognitive functioning.
Change in overall cognitive functioning | Baseline and 18 Months
  As measured by the difference between the Montreal Cognitive Assessment (MoCA) score at baseline and at 18-months follow-up.The MoCA measures eight domains commonly affected by mild cognitive impairment. The one-page 30-point test includes assessments of short-term and delayed memory recall, visuospatial abilities, language, orientation to time and space, and executive functions including attention, concentration, and working memory. The MoCA has been shown to be sensitive to change over time. Scores on the MocA range from 0-30 with higher scores indicating better cognitive functioning.
Attention/working memory at baseline as measured by the Trail Making A Test | Baseline
  The Trail Making Test is a quickly and easily administered test which assesses cognitive abilities such as visual-conceptual and visual-motor tracking, sustained attention, and task alternation abilities. Administration time for the Trail Making Test A is 5 minutes.
Attention/working memory change from baseline to 18-months follow-up as measured by the Trail Making A Test | 18 months
  The Trail Making Test is a quickly and easily administered test which assesses cognitive abilities such as visual-conceptual and visual-motor tracking, sustained attention, and task alternation abilities. Administration time for the Trail Making Test A is 5 minutes.
Attention/working memory at baseline as measured by the Symbol Digit Modalities Test (SDMT) | Baseline
  Symbol Digit Modalities Test (SDMT) takes five minutes to complete and has demonstrated sensitivity in detecting changes in cognitive functioning over time.
Attention/working memory change from baseline to 18-months follow-up as measured by the Symbol Digit Modalities Test | Baseline and 18- months follow-up
  Symbol Digit Modalities Test (SDMT) takes five minutes to complete and has demonstrated sensitivity in detecting changes in cognitive functioning over time.
Executive function at baseline as measured by the Clock Drawing Test | Baseline
  The Clock Drawing Test is a quick screening test for cognitive dysfunction secondary to a range of neurological disorders and takes less than 5 minutes to administer.
Executive function change from baseline to 18-months follow-up as measured by the Clock Drawing Test | Baseline and 18-month follow-up
  The Clock Drawing Test is a quick screening test for cognitive dysfunction secondary to a range of neurological disorders and takes less than 5 minutes to administer.
Executive function at baseline as measured by the Trail Making Test B | Baseline
  The Trail Making Test is a quickly and easily administered test which assesses cognitive abilities such as visual-conceptual and visual-motor tracking, sustained attention, and task alternation abilities. Administration time for the Trail Making Test B is 10 minutes.
Executive function change from baseline to 18-months follow-up as measured by the Trail Making Test B | Baseline and 18-month follow-up
  The Trail Making Test is a quickly and easily administered test which assesses cognitive abilities such as visual-conceptual and visual-motor tracking, sustained attention, and task alternation abilities. Administration time for the Trail Making Test B is 10 minutes.
Language at baseline as measured by the Animal Naming Test | Baseline
  The Animal Naming Test is a semantic fluency test that takes one minute to administer.
Language change from baseline to 18-month follow-up as measured by the Animal Naming Test | Baseline and 18-months follow-up
  The Animal Naming Test is a semantic fluency test that takes one minute to administer.
Language at baseline as measured by the Boston Naming Test | Baseline
  The Boston Naming Test measures confrontational word retrieval and takes about 15 minutes to administer.
Language change from baseline to 18-months follow-up as measured by the Boston Naming Test | Baseline and 18-months follow-up
  The Boston Naming Test measures confrontational word retrieval and takes about 15 minutes to administer.
Language change between baseline and 18-month follow-up as measured by the Boston Naming Test | Baseline
  The Boston Naming Test measures confrontational word retrieval and takes about 15 minutes to administer.
Memory at baseline as measured by the Free and Cued Selective Reminding Test | Baseline
  The Free and Cued Selective Reminding Test is an episodic memory test which assesses immediate and delayed free and cued-facilitated recall.
Memory change from baseline to 18-months follow-up as measured by the Free and Cued Selective Reminding Test | Baseline and 18-months follow-up
  The Free and Cued Selective Reminding Test is an episodic memory test which assesses immediate and delayed free and cued-facilitated recall.
Memory at baseline as measured by the Brief Visuospatial Memory Test-Revised Selective Reminding Test | Baseline
  The Brief Visuospatial Memory Test-Revised is a brief measure of visuospatial memory that takes approximately 45 minutes to administer.
Memory change from baseline to 18-months follow-up as measured by the Brief Visuospatial Memory Test-Revised | Baseline and 18-months follow-up
  The Brief Visuospatial Memory Test-Revised is a brief measure of visuospatial memory that takes approximately 45 minutes to administer.
Memory change between baseline and 18-month follow-up | Baseline and 18-month follow-up
  As measured by the change in Free and Cued Selective Reminding Test and the Brief Visuospatial Memory Test-Revised scores at baseline and at 18-months follow-up.
Visuospatial at baseline as measured by the Judgement of Line Orientation Test | Baseline
  Judgement of Line Orientation measures visuospatial perception and takes less than 15 minutes to administer.
Visuospatial change from baseline to 18-months follow-up as measured by the Judgement of Line Orientation Test | Baseline and 18-months follow-up
  Judgement of Line Orientation measures visuospatial perception and takes less than 15 minutes to administer.
Visuospatial at baseline as measured by the Intersecting Pentagons Test | Baseline
  Intersecting Pentagons is a measure of visuospatial sense that takes less than 5 minutes to administer.
Visuospatial change from baseline to 18-months follow-up as measured by the Intersecting Pentagons Test | Baseline and 18-months follow-up
  Intersecting Pentagons is a measure of visuospatial perception that takes less than 5 minutes to administer.
Estrogen levels in blood at baseline | Baseline
  Estrogen levels (picograms of estradiol per milliliter of serum) will be measured via blood draw performed at baseline
Progesterone levels in blood as baseline | Baseline
  Progesterone levels (nanograms of progesterone per milliliter of serum) will be measured via blood draw at baseline
Testosterone levels in blood at baseline | Baseline
  Levels of free testosterone (picograms testosterone per milliliter serum) and total testosterone (nanograms testosterone/deciliter serum) will be measured via blood draw performed at the baseline visit.

SECONDARY OUTCOMES:
Cholinergic terminal binding potential at baseline | Baseline
  Measured by PFC [18F]VAT VT and BPND
Cholinergic terminal binding potential change between baseline and 18-months follow-up | Baseline and 18-month follow-up
  Measured by PFC [18F]VAT VT and BPND
MRI Fractional anisotropy (FA) Values at baseline | Baseline
  As measured by fMRI at baseline
Change in MRI Fractional anisotropy (FA) Values from baseline to 18-months follow-up | Baseline and 18-months follow-up
  As measured by fMRI at baseline and 18-months follow-up
MRI Resting-state functional connectivity at baseline | Baseline
  As measured by fMRI
MRI Resting-state functional connectivity change between baseline and 18-months follow-up | Baseline and 18-months follow-up
  As measured by fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Huang, PhD, Principal Investigator — Stony Brook Medical Center; Carine Maurer, PhD, Principal Investigator — Stony Brook Medical Center
Locations (1):
- Stony Brook Medical Center, Stony Brook, New York, United States